CLINICAL TRIAL: NCT01162187
Title: Secondary Prevention in Acute Coronary Syndromes: Long-term Survival in Relation to the Number and Combination of Evidence-based Therapies Prescribed Prior to Discharge (a CALIBER Study)
Brief Title: Secondary Prevention in Acute Coronary Syndromes: A CALIBER Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Barts & The London NHS Trust (Other); University of Leicester (Other)
Responsible Party: Dr Owen Nicholas, University College London
Other Study IDs: CALIBER-09-02
Record Dates: First submitted 2010-07-01; First posted 2010-07-14 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: Acute Coronary Syndrome
Keywords: secondary prevention; aspirin; beta blocker; ACE inhibitor; statin; acute coronary syndrome; myocardial infarction; unstable angina; trends
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
All contemporary guidelines for secondary prevention in acute coronary syndromes recommend a combination of aspirin, beta-blockers, ACE-inhibitors and statins. Yet underutilisation of these drugs is common. We do not know in detail what drives underutilisation, nor what its long term consequences are for survival after discharge from hospital. Also unknown is whether potential adverse effects of underutilisation are the same for individual secondary prevention drugs.

This study will assess the impact of secondary prevention underutilisation on survival.

DETAILED DESCRIPTION:
Using information from an England and Wales audit of acute coronary syndromes (the Myocardial Ischaemia National Audit Project (MINAP)) we aim to assess:

(i) Survival from first time MINAP-registered event to death as a function of secondary prevention medications: To what degree do the effects of medications (assumed equal, independent and additive) relate to patient survival? Is there evidence of a differential effect of discharge medications? (ii) (a) Survival from first time MINAP-registered event to death or second time MINAP-registered event as a function of secondary prevention medications: To what degree do the effects of medications (assumed equal, independent and additive) relate to competing risks? Is there evidence of a differential effect of discharge medications? (b) Survival from first time MINAP-registered event to death or second time MINAP-registered phenotyped as STEMI, NSTEMI or Unstable Angina. To what degree do the effects of medications (assumed equal, independent and additive) relate to competing risks? Is there evidence of a differential effect of discharge medications? (iii) What impact would ensuring all medication is taken have on event free survival?

This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the NIHR and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (GPRD) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Acute Coronary Syndrome who have been registered with the MINAP database.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with data entered into the Myocardial Ischaemia National Audit Project (MINAP) database in England and Wales.
Sampling Method: Non-Probability Sample
Enrollment: 400000 (Estimated)
Dates: Start 2003-07; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | Due to follow up an average of 3 years.
  Mortality as tracked by the Office for National Statistics

SECONDARY OUTCOMES:
Competing risks between acute coronary syndrome phenotypes | Due to follow up an average of 3 years.
  Stable Angina, Unstable Angina, STEMI and NSTEMI will be treated both as startpoints and endpoints in transitions between phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Owen M Nicholas, PhD, Principal Investigator — University College, London

REFERENCES:
- [Background] National Collaborating Centre for Primary Care (UK). Post Myocardial Infarction: Secondary Prevention in Primary and Secondary Care for Patients Following a Myocardial Infarction [Internet]. London: Royal College of General Practitioners (UK); 2007 May. Available from http://www.ncbi.nlm.nih.gov/books/NBK49343/ PMID 21290635
- [Background] Goodman SG, Huang W, Yan AT, Budaj A, Kennelly BM, Gore JM, Fox KA, Goldberg RJ, Anderson FA Jr; Expanded Global Registry of Acute Coronary Events (GRACE2) Investigators. The expanded Global Registry of Acute Coronary Events: baseline characteristics, management practices, and hospital outcomes of patients with acute coronary syndromes. Am Heart J. 2009 Aug;158(2):193-201.e1-5. doi: 10.1016/j.ahj.2009.06.003. PMID 19619694
- [Background] Chew DP, Anderson FA, Avezum A, Eagle KA, FitzGerald G, Gore JM, Dedrick R, Brieger D; GRACE Investigators. Six-month survival benefits associated with clinical guideline recommendations in acute coronary syndromes. Heart. 2010 Aug;96(15):1201-6. doi: 10.1136/hrt.2009.184853. Epub 2010 Jun 7. PMID 20530127
- [Background] Bramlage P, Messer C, Bitterlich N, Pohlmann C, Cuneo A, Stammwitz E, Tebbenjohanns J, Gohlke H, Senges J, Tebbe U. The effect of optimal medical therapy on 1-year mortality after acute myocardial infarction. Heart. 2010 Apr;96(8):604-9. doi: 10.1136/hrt.2009.188607. Epub 2010 Mar 29. PMID 20353936
- See also: CALIBER is based on linking the national myocardial infarction register to the rich longitudinal primary care record — http://www.caliberresearch.org/